CLINICAL TRIAL: NCT03565445
Title: A Phase 1b Study of ASP1948, Targeting an Immune Modulatory Receptor as a Single Agent and in Combination With a PD-l Inhibitor (Nivolumab or Pembrolizumab) in Subjects With Advanced Solid Tumors
Brief Title: A Study of ASP1948, Targeting an Immune Modulatory Receptor as a Single Agent and in Combination With a PD-l Inhibitor (Nivolumab or Pembrolizumab) in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1948-CL-0101; 2018-003873-82 (EudraCT Number); KEYNOTE-A87 (Other: Merck); jRCT2031200341 (Registry Identifier: Japan Registry for Clinical Trials (jRCT)); MK-3475-A87 (Other: Merck)
Record Dates: First submitted 2018-05-25; First posted 2018-06-21 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors
Keywords: NSCLC; Tumors; squamous cell carcinoma of the head and neck (SCCHN); Oncology; breast cancer; ASP1948; mCRPC; ovarian cancer; Locally advanced or metastatic solid tumor malignancies; pancreatic cancer; Advanced solid tumors
MeSH Terms: conditions — Neoplasms; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- ASP1948 70 mg Monotherapy Dose Escalation (Experimental): Participants have received ASP1948 70 mg intravenously, on day 1 of every 2-week (Q2W) cycle for a period of up to 24 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948
- ASP1948 200 mg Monotherapy Dose Escalation (Experimental): Participants have received ASP1948 200 mg intravenously, on day 1 of Q2W cycle for a period of up to 24 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948
- ASP1948 700 mg Monotherapy Dose Escalation (Experimental): Participants have received ASP1948 700 mg intravenously, on day 1 of every 2 week cycle for a period of up to 24 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948
- ASP1948 1200 mg Monotherapy Dose Expansion (Experimental): Participants have received ASP1948 1200 mg intravenously, on day 1 of every 2 week cycle for a period of up to 24 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948
- ASP1948 2000 mg Monotherapy Dose Escalation (Experimental): Participants have received ASP1948 2000 mg intravenously, on day 1 of every 2 week cycle for a period of up to 24 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948
- ASP1948 3000 mg Monotherapy Dose Escalation (Experimental): Participants have received ASP1948 3000 mg intravenously, on day 1 of every 3-week (Q3W) cycle for a period of up to 16 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received treatment for an additional 16 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948
- ASP1948 2000 mg Monotherapy Dose Expansion (Experimental): Participants have received ASP1948 2000 mg intravenously, on day 1 of Q2W cycle for a period of up to 24 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948
- ASP1948 1200 mg + Nivolumab 240 mg CT Dose Escalation (Experimental): Participants have received ASP1948 1200 mg intravenously in combination with nivolumab 240 mg administered as a 30 minute intravenous infusion, on day 1 of Q2W cycle for a period of up to 24 cycles or until a discontinuation criterion is met. Qualifying participants have entered a re-treatment period and have received combination treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948; Drug: nivolumab
- ASP1948 2000 mg+ Nivolumab 240 mg CT Dose Escalation (Experimental): Participants have received ASP1948 2000 mg intravenously in combination with nivolumab 240 mg administered as a 30 minute intravenous infusion, on day 1 of Q2W cycle for a period of up to 24 cycles or until a discontinuation criterion is met. Qualifying participants have entered a re-treatment period and have received combination treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948; Drug: nivolumab
- ASP1948 2000 mg + Nivolumab 240 mg CT Dose Expansion (Experimental): Participants have received ASP1948 2000 mg intravenously in combination with nivolumab 240 mg administered as a 30 minute intravenous infusion, on day 1 of every 2 week cycle for a period of up to 24 cycles or until a discontinuation criterion is met. Qualifying participants have entered a re-treatment period and have received combination treatment for an additional 24 cycles or until a discontinuation criteria is met.
  Interventions: Drug: ASP1948; Drug: nivolumab
- ASP1948 2000 mg + Pembrolizumab 400 mg CT Dose Escalation (Experimental): Participants have received ASP1948 2000 mg intravenously on day 1 of Q2W cycle in combination with pembrolizumab 400 mg administered as a 30 minute intravenous infusion, on day 1, once every 6 weeks (Q6W) for a period of up to 24 cycles or until a discontinuation criterion is met. Qualifying participants have entered a re-treatment period and have received combination treatment for an additional 24 cycles or until a discontinuation criteria is met. Participants who completed 24 cycles of treatment and have entered the follow-up period with PR or SD are allowed to continue on pembrolizumab alone for a period of up to an additional 10 doses of pembrolizumab. If the participant is eligible for a re-treatment period during follow up, administration of pembrolizumab alone is discontinued and combination therapy with ASP1948 is resumed per the protocol.
  Interventions: Drug: ASP1948; Drug: pembrolizumab
- ASP1948 3000 mg + Pembrolizumab 200 mg CT Dose Escalation (Experimental): Participants have received ASP1948 3000 mg intravenously in combination with pembrolizumab 200 mg administered as a 30 minute intravenous infusion, on day 1 of Q3W cycle for a period of up to 16 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received combination treatment for an additional 16 cycles or until a discontinuation criteria is met. Participants who completed 16 cycles of treatment and have entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant is eligible for a re-treatment period during follow up, administration of pembrolizumab alone is discontinued and combination therapy with ASP1948 is resumed per the protocol.
  Interventions: Drug: ASP1948; Drug: pembrolizumab
- ASP1948 3000 mg + Pembrolizumab 200 mg CT Dose Expansion (Experimental): Participants have received ASP1948 3000 mg intravenously in combination with pembrolizumab 200 mg administered as a 30 minute intravenous infusion, on day 1 of Q3W cycle for a period of up to 16 cycles or until a discontinuation criterion is met during treatment period. Qualifying participants have entered a re-treatment period and have received combination treatment for an additional 16 cycles or until a discontinuation criteria is met. Participants who completed 16 cycles of treatment and have entered the follow-up period with PR or SD were allowed to continue on pembrolizumab alone for a period of up to an additional 19 cycles. If the participant is eligible for a re-treatment period during follow up, administration of pembrolizumab alone is discontinued and combination therapy with ASP1948 is resumed per the protocol.
  Interventions: Drug: ASP1948; Drug: pembrolizumab

INTERVENTIONS:
Drug: ASP1948 — Intravenously (IV)
Drug: nivolumab — Intravenously (IV)
  Arms: ASP1948 1200 mg + Nivolumab 240 mg CT Dose Escalation; ASP1948 2000 mg + Nivolumab 240 mg CT Dose Expansion; ASP1948 2000 mg+ Nivolumab 240 mg CT Dose Escalation
Drug: pembrolizumab — Intravenously (IV)
  Other Names: KEYTRUDA®
  Arms: ASP1948 2000 mg + Pembrolizumab 400 mg CT Dose Escalation; ASP1948 3000 mg + Pembrolizumab 200 mg CT Dose Escalation; ASP1948 3000 mg + Pembrolizumab 200 mg CT Dose Expansion

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety profile of ASP1948 when administered as a single agent and in combination with nivolumab or pembrolizumab in participants with locally advanced (unresectable) or metastatic solid tumors; characterize the pharmacokinetic profile of ASP1948 when administered as a single agent and in combination with nivolumab or pembrolizumab and determine the recommended Phase 2 dose (RP2D) of ASP1948 when administered as a single agent and in combination with nivolumab or pembrolizumab. This study will also evaluate the antitumor effect of ASP1948 when administered as a single agent and in combination with nivolumab or pembrolizumab.

DETAILED DESCRIPTION:
This is a dose-escalation and expansion study of ASP1948 as a single agent and in combination with nivolumab or pembrolizumab. The study consists of 3 periods for monotherapy and combination therapy: screening, treatment and follow up, followed by an optional Re-treatment period for participants that qualify.

The escalation cohorts will evaluate escalating dose levels of ASP1948 in participants with locally advanced (unresectable) or metastatic solid tumor malignancies.

After discontinuation of study drug, all participants will complete an end-of-treatment visit, along with 30-day and 90-day safety follow-up visits from the last dose of study drug.

For dose expansion, the tumor-specific cohorts will include participants with squamous cell carcinoma of the head and neck (SCCHN), non-small cell lung cancer (NSCLC), metastatic castration-resistant prostate cancer (mCRPC), ovarian cancer, pancreatic cancer and breast cancer, as well as any tumor types that respond to study drug treatment during dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has locally-advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) that is confirmed by available pathology records or current biopsy, and has received all standard therapies (unless the therapy is contraindicated or intolerable) felt to provide clinical benefit.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1.
* Subject's last dose of prior antineoplastic therapy, including any immunotherapy, was at least 21 days prior to initiation of study drug administration. A subject with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutation-positive NSCLC is allowed to remain on EGFR tyrosine kinase inhibitor (TKI) or ALK inhibitor therapy until 4 days prior to the start of study drug administration.
* Subject has completed any radiotherapy (including stereotactic radiosurgery) at least 14 days prior to study drug administration.
* Subject with metastatic castration-resistant prostate cancer (mCRPC) (positive scan and/or soft tissue disease documented by computed tomography/magnetic resonance imaging) meets both of the following:

  * Subject has serum testosterone ≤ 50 ng/dL at screening.
  * Subject has had an orchiectomy or plans to continue androgen deprivation therapy (ADT) for the duration of study treatment.
* Subject has adequate organ function as indicated by laboratory values. (If a subject has received a recent blood transfusion, the laboratory tests must be obtained ≥ 28 days after any blood transfusion.) Subjects can be on a stable dose of erythropoietin (≥ approximately 3 months). Note: Growth factors, colony stimulating factors are not permitted in the screening period.
* Female subject must either:

  * Be of non-childbearing potential: post-menopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or; documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy).
  * Or, if of childbearing potential: Agree not to try to become pregnant during the study treatment and for 6 months after the final study drug administration; and have a negative urine or serum pregnancy test prior to study drug administration; and if heterosexually active, agree to consistently use 1 form of highly effective birth control starting at screening and throughout the study treatment and 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study treatment, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study treatment, and for 6 months after the final study drug administration.
* A sexually active male subject with female partner(s) who are of childbearing potential is eligible if :

  * The male subject agrees to use a male condom starting at screening and continues throughout the study treatment, and for 6 months after the final study drug administration.
  * The male subject has not had a vasectomy or is not sterile, as defined below and the subject's female partner(s) is utilizing 1 form of highly effective birth control starting at screening and continuing throughout the study treatment and for 6 months after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study treatment, and for 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study treatment and for 6 months after the final study drug administration.
* Subject agrees not to participate in another interventional study while receiving study drug (subjects who are currently in the follow-up period of an interventional clinical trial are allowed).

Additional Inclusion Criteria for Subjects in the Expansion Cohorts:

* Subject has at least 1 measurable lesion per RECIST 1.1. The measureable lesion must be outside the field of radiation if subject had prior radiotherapy. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Subjects with mCRPC who do not have measurable lesions must have at least 1 of the following:

  * Progression with 2 or more new bone lesions, or
  * Prostate specific antigen (PSA) progression (defined as a minimum of 3 rising PSA levels with an interval of ≥ 1 week between each determination) within 6 weeks prior to study drug administration and a PSA value at the screening visit ≥ 2 ng/mL.
* Subject consents to provide available tumor specimen in a tissue block or unstained serial slides obtained within 8 to 56 days prior to first dose of study treatment. Note: This does not apply to subjects with mCRPC who do not have measurable disease.
* Subject is an appropriate candidate for tumor biopsy and consents to undergoing a tumor biopsy (core needle biopsy or excision) during the treatment period. Note: This does not apply to subjects with mCRPC who do not have measurable disease.
* Subject meets one of the following:

  * Subject has the tumor type for which a confirmed response was observed in a monotherapy or in combination with nivolumab dose escalation or RP2D cohort; or
  * ASP1948 monotherapy or in combination with pembrolizumab expansion cohort is opened due to achieving predicted efficacious exposure, subject has squamous cell carcinoma of the head and neck (SCCHN); or
  * RP2D monotherapy cohort is opened and subject has NSCLC, mCRPC, ovarian cancer, pancreatic cancer or breast cancer; or
  * RP2D combination with pembrolizumab expansion cohort, is opened and subject has NSCLC (all PD-L1 status), NSCLC PD-L1 high*, ovarian cancer, colorectal cancer, or breast cancer.

    * NSCLC with PD-L1 high expressing tumor as determined by immunohistochemistry at a central laboratory during the screening period.

Additional Inclusion Criteria for Re-treatment:

Subjects may be eligible for study drug re-treatment if the study remains open and the subject continues to meet all of the eligibility criteria above (except prior use of this drug) and the following conditions:

* Subject stopped initial treatment with ASP1948 or ASP1948 in combination with nivolumab or pembrolizumab after attaining a confirmed CR or PR or SD.
* Subject experienced a confirmed disease progression by iRECIST (iCPD) after stopping their initial treatment with ASP1948 or ASP1948 in combination with nivolumab or pembrolizumab.
* Subject did not receive any prohibited anti-cancer treatment since the last dose of ASP1948 or ASP1948 in combination with nivolumab or pembrolizumab.
* Subject did not experience a toxicity that met the discontinuation criteria during the initial treatment with ASP1948 or ASP1948 in combination with nivolumab or pembrolizumab.

Exclusion Criteria:

* Subject weighs < 45 kg.
* Subject has received investigational therapy (other than an investigational epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) in a subject with EGFR mutations or ALK inhibitor in a subject with an ALK mutation) within 21 days prior to start of study drug.
* Subject requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to study drug administration. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent(defined as up to 30 mg per day of hydrocortisone, 2 mg per day of dexamethasone or up to 10 mg per day of prednisone) are allowed. Note: Corticosteroids for prophylaxis (e.g., contrast dye allergy) or for brief treatment of conditions not related to study treatment (e.g., delayed-type hypersensitivity reaction caused by a contact allergen) is also allowed.
* Subject has symptomatic central nervous system (CNS) metastases or subject has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Subjects with previously treated CNS metastases are eligible, if the subject is clinically stable and has no evidence of CNS progression by imaging for at least 28 days prior to start of study treatment and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone, > 2 mg per day of dexamethasone or > 10 mg per day of prednisone or equivalent) for longer than 14 days.
* Subject has leptomeningeal disease as a manifestation of the current malignancy.
* Subject has an active autoimmune disease that has required systemic treatment in the past 2 years. Subjects with type 1 diabetes mellitus, stable endocrinopathies maintained on appropriate replacement therapy and skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment are allowed.
* Subject was discontinued from prior immunomodulatory therapy due to a Grade ≥ 3 toxicity that was mechanistically related (e.g., immune related) to the agent.
* Subject has known history of serious hypersensitivity reaction to a known ingredient of ASP1948, nivolumab or pembrolizumab or severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Subject with positive Hepatitis B virus antibodies and surface antigen (indicating acute Hepatitis B virus (HBV) or chronic HBV) or Hepatitis C (HCV ribonucleic acid (RNA) [(qualitative or quantitative)]. Hepatitis C RNA testing is not required in subjects with negative Hepatitis C antibody testing. Hepatitis B virus antibodies are not required in subjects with negative Hepatitis B surface antigen.
* Subject has received a live vaccine against infectious diseases within 28 days prior to initiation of study treatment.
* Subject has a history of drug-induced pneumonitis (interstitial lung disease), a history of (non-infectious) pneumonitis that required steroids, radiation pneumonitis or currently has pneumonitis.
* Subject has an active infection requiring systemic therapy within 14 days prior to study drug treatment.
* Subject is expected to require another form of antineoplastic therapy while on study treatment.
* Subject has an uncontrolled intercurrent illness including, but not limited to cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject's AEs (excluding alopecia) from prior therapy have not improved to Grade 1 or baseline within 14 days prior to start of study treatment.
* Subject has significant cardiovascular disease including:

  * Subject has inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
  * Subject has a history of myocardial infarction or unstable angina within 6 months prior to day 1.
  * Subject has New York Heart Association Class II or greater chronic heart failure (CHF).
  * History of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to study treatment.
  * Subject has significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study treatment.
* Subject has a history of hemoptysis (bright red blood of ½ teaspoon or more per episode) within 12 weeks prior to study treatment.
* Subject has evidence of a bleeding diathesis or significant coagulopathy.
* Subject has inadequate recovery from prior surgical procedure or has had a major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to day 1, or anticipates the need for a major surgical procedure during the course of the study or minor surgery within 7 days of starting study treatment.
* Subject has initiated new treatment with medications that affect the coagulation cascade with an international normalized ratio (INR) ≥ 2 such as vitamin K antagonists, heparins and direct thrombin inhibitors or the use of factor Xa inhibitors within 28 days prior to the start of study treatment. Note: If the subject started receiving such medications more than 28 days prior to the start of study treatment and needs to continue, this is allowed. However, new anticoagulation may not be initiated within 28 days prior to the start of study treatment.
* Subject has any condition that makes the subject unsuitable for study participation.
* Subject has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
* Subject has had an allogeneic tissue solid organ transplant.
* Subject has known history of COVID-19 positive polymerase chain reaction (PCR) test within 4 weeks prior to start of study treatment.

Additional Exclusion Criteria for Subjects in Expansion Cohorts:

* Subject has a prior malignancy active (i.e., requiring treatment or intervention) within the previous 2 years, except for locally curable malignancies that have been apparently cured, which are allowed, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
* Subject has received prior treatment with a neuropilin-1 (NRP1) inhibitor.

Additional Exclusion Criteria for Re-treatment:

* Subjects who have completed 40 weeks (ASP1948 monotherapy or combination therapy with nivolumab cohorts) or 57 weeks (ASP1948 combination therapy with pembrolizumab) of follow-up with disease control are not eligible for retreatment.
* Subject currently has an ongoing Adverse Event (AE) related to the initial ASP1948 or ASP1948 in combination with nivolumab or pembrolizumab treatment that meets the criteria for treatment interruption or discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  DLT is any AE that cannot be attributed to a cause other than study drug:
  Grade (Gr) 4 NTP or Gr ≥ 3 febrile NTP Gr 4 TCP; or Gr 3 TCP accompanied by bleeding that requires transfusion Gr 4 anemia or Gr 3 anemia requiring transfusion Gr ≥ 3 NHAE Gr ≥ 2 pneumonitis AST or ALT > 5x upper limit of normal (ULN; Gr ≥ 3) without liver metastases AST or ALT > 8 x ULN in participants with liver metastases AST or ALT > 3 x ULN & total bilirubin > 2 x ULN (in participant with Gilbert syndrome: AST or ALT > 3x ULN & direct bilirubin > 1.5 x ULN) Total bilirubin > 3x ULN (Gr ≥ 3) Gr ≥ 2 encephalopathy, meningitis, or motor or sensory neuropathy Gr ≥ 2 pulmonary or CNS hemorrhage Gr ≥ 3 hemorrhage GBS or MS/MG IRR leading to infusion discontinuation Prolonged delay in initiating cycle 2 due to TRT Any TRT that caused participant to discontinue treatment during DLT period Missing >25% of ASP1948 or pembrolizumab doses as a result of drug-related AE(s) during DLT period Gr 5 toxicity.
Number of Participants with Adverse Events (AEs) | From first dose until 90 days after last dose (up to 823 days)
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An AE is considered "serious" if, it resulted in any of the following outcomes: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly, or birth defect; requires inpatient hospitalization; or leads to prolongation of hospitalization; other medically important events. TEAE is defined as an AE observed after starting administration of the study drug.
Number of Participants with Immune-related AEs | From first dose until 30 days after last dose (up to 763 days)
  Immune-related AEs observed with currently approved checkpoint inhibitors (CPIs) include rash, oral mucositis, dry mouth, colitis/diarrhea, hepatitis, pneumonitis, and endocrinopathies (hypophysitis, hypothyroidism, hyperthyroidism, adrenal insufficiency and Type 1 diabetes mellitus). Other less frequent irAEs associated with CPIs include: nephritis; pancreatitis; myositis; arthritis; neurologic toxicities (Guillain-Barre syndrome, myasthenia gravis, posterior reversible encephalopathy syndrome, aseptic meningitis, enteric neuropathy, transverse myelitis, and autoimmune encephalitis), cardiotoxicity (myocarditis and conduction abnormalities); hematologic toxicity (red cell aplasia, neutropenia, thrombo-cytopenia, acquired hemophilia A, and cryoglobulinemia); and eye inflammation (episcleritis, conjunctivitis, uveitis or orbital inflammation). TEAE is defined as an AE observed after starting administration of the study drug.
Number of Participants with Eastern Cooperative Oncology Group (ECOG) performance status | End of Treatment (Baseline up to 733 days)
  The ECOG is used to assess performance status. Number of participants in each of the ECOG PS grade were reported.
  0 = Fully active, able to carry on all predisease performance without restriction;
  1. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature;
  2. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours;
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours;
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  Negative change scores indicate an improvement. Positive scores indicate a decline in performance.
Pharmacokinetics (PK) of ASP1948 (Cycle 1): Area Under The Concentration-Time Curve From The Time Zero to The Last Measurable Concentration (AUClast) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  AUClast is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): AUClast | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  AUClast is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Area Under the Concentration-Time Curve From the Time of Dosing Extrapolated to Time Infinity (AUCinf) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  AUCinf is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Percentage of AUCinf Due to Extrapolation From Time of The Last Measurable Concentration To Time Infinity (AUCinf %extrap) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  AUCinf %extrap is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Area Under The Concentration-Time Curve From The Time of Dosing to The Start of Next Dosing Interval (AUCtau) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  AUCtau is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Maximum Concentration (Cmax) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  Cmax is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): Cmax | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  Cmax is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): Trough Concentration (Ctrough) | Cycle 10: Predose
  Ctrough is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Time of The Maximum Concentration (tmax) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  tmax is derived from the PK serum samples collected
PK of ASP1948 (Cycle 10): tmax | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  tmax is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): AUCtau | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  AUCtau is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Terminal Elimination Half-Life ( t1/2) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  t1/2 is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Time of Last Measurable Concentration (tlast) | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  tlast is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): Terminal Elimination Half-Life ( t1/2) | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  t1/2 is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): tlast | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  tlast is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Total Clearance (CL) after Intravenous Dosing | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  CL is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): CL after Intravenous Dosing | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  CL is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Volume of Distribution During the Terminal Elimination Phase (Vz) After Intravenous Dosing | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  Vz is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): Vz After Intravenous Dosing | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  Vz is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 1): Apparent Volume of Distribution at Steady State (Vss) after Intravenous Dosing | Cycle 1: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  Vss is derived from the PK serum samples collected.
PK of ASP1948 (Cycle 10): Vss After Intravenous Dosing | Cycle 10: pre-dose, within 20 minutes after end of dosing, 4 hours, 24 hours, 48 hours, 168 hours post dose
  Vss is derived from the PK serum samples collected.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as per RECIST V1.1 | From start of study until radiographical progression or date of censoring (maximum treatment duration: up to 733 days)
  ORR as per RECIST 1.1 is defined as the percentage of participants for each dose level whose best overall response is rated as confirmed CR or PR. CR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR is defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
ORR as per iRECIST V1.1 | From start of study until radiographical progression or date of censoring (maximum treatment duration: up to 733 days)
  ORR as per iRECIST is defined as the percentage of participants for each dose level whose best overall response is rated as confirmed iCR or iPR. iCR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR is defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Duration of Response (DOR) as per RECIST V1.1 | From the date of the first response CR/PR to the date of radiographical progression or date of censoring (maximum treatment duration: up to 733 days)
  DOR as per RECIST 1.1 is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression or date of censoring. CR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR is defined as at least a 30% decrease in the sum of diameters (longest for non nodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
DOR as per iRECIST | From the date of the first response CR/PR to the date of radiographical progression or date of censoring (maximum treatment duration: up to 733 days)
  DOR as per iRECIST is defined as the time from the date of the first response iCR/iPR (whichever is first recorded) to the date of radiographical progression or date of censoring. iCR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR is defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Persistence of response after discontinuation per RECIST V1.1 | From date of treatment discontinuation to the date of radiographical progression or date of censoring (maximum duration: up to 733 days)
  Persistence of response as per RECIST 1.1 is defined as the time from the date of treatment discontinuation to the date of radiographical progression or date of censoring. Persistence of response is derived for participants who at the time of treatment discontinuation had a confirmed response of CR or PR based on RECIST 1.1. CR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR is defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Persistence of response after discontinuation per iRECIST | From date of treatment discontinuation to the date of radiographical progression or date of censoring (maximum treatment duration: up to 733 days)
  Persistence of response as per iRECIST is defined as the time from the date of treatment discontinuation to the date of radiographical progression or date of censoring. Persistence of response is derived for participants who at the time of treatment discontinuation had a confirmed response of iCR or iPR. iCR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. iPR is defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Disease Control Rate (DCR) by RECIST 1.1 | From start of study until radiographical progression or date of censoring (maximum treatment duration: up to 733 days)
  DCR as per RECIST 1.1 is defined as percentage of participants for each dose level whose BOR is rated as confirmed CR, PR or Stable Disease (SD). CR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR is defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD is defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters. Progressive disease (PD): >= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression.
DCR by iRECIST | From start of study until radiographical progression or date of censoring (maximum treatment duration: up to 733 days)
  DCR as per RECIST 1.1 is defined as percentage of participants for each dose level whose BOR is rated as confirmed CR, PR or Stable Disease (SD). CR is defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR is defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD is defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters. Progressive disease (PD): >= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (42):
- United States (17):
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Norton Cancer Institute, Louisville, Kentucky
  - Cancer Center at Greater Baltimore Medical, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - UPMC- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute - SCRI, Nashville, Tennessee
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Virginia Cancer Care Specialist, PC, Fairfax, Virginia
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
- Canada (2):
  - Site CA15002, Edmonton
  - Site CA15004, Montreal
- Italy (2):
  - Site IT39008, Milan
  - Site IT39006, Modena
- Japan (2):
  - Site JP81002, Chiba
  - Site JP81001, Tokyo
- Site PT35104, Porto, Portugal
- South Korea (7):
  - Site KR82001, Seoul
  - Site KR82002, Seoul
  - Site KR82003, Seoul
  - Site KR82004, Seoul
  - Site KR82005, Seoul
  - Site KR82006, Seoul
  - Site KR82007, Seoul
- Spain (8):
  - Site ES34002, Barcelona
  - Site ES34006, Barcelona
  - Site ES34010, Barcelona
  - Site ES34014, Barcelona
  - Site ES34003, Cataluna
  - Site ES34004, Cataluna
  - Site ES34007, Madrid
  - Site ES34012, Madrid
- Taiwan (2):
  - Site TW88601, Taipei
  - Site TW88602, Taipei
- Site GB44006, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Bao R, Surriga O, Olson DJ, Allred JB, Strand CA, Zha Y, Carll T, Labadie BW, Bastos BR, Butler M, Hogg D, Musi E, Ambrosini G, Munster P, Schwartz GK, Luke JJ. Transcriptional analysis of metastatic uveal melanoma survival nominates NRP1 as a therapeutic target. Melanoma Res. 2021 Feb 1;31(1):27-37. doi: 10.1097/CMR.0000000000000701. PMID 33170593
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14538&tenant=MT_AST_9011